CLINICAL TRIAL: NCT02727283
Title: A Phase 1, Randomized, Placebo-Controlled, Double-Blind, Ascending Dose Escalating, 4 Period Crossover Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Food Effect of Single Doses of GSK3179106, a REarranged During Transfection (RET) Growth Factor Receptor Tyrosine Kinase Inhibitor, in Normal Healthy Volunteers
Brief Title: A Phase 1, Randomized, Placebo-Controlled, Ascending Cohort, Dose Escalation Study in Normal Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 204729
Record Dates: First submitted 2015-12-14; First posted 2016-04-04 (Estimated); Last update posted 2017-05-08 (Actual); Status verified 2017-05

CONDITIONS: Irritable Bowel Syndrome
Keywords: Healthy volunteer; Safety; Pharmacokinetics; Dose escalation; GSK3179106; Rearranged during Transfection; Irritable Bowel Syndrome; Adults
MeSH Terms: conditions — Irritable Bowel Syndrome; Multiple Endocrine Neoplasia Type 2a

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort 1 (Experimental): Subjects will receive 1 placebo and 3 escalating doses in one of the four treatment periods. The planned dose range is 10 mg to 200 mg. A review of safety and tolerability will occur prior to administration of the next dose level and the same procedure will be followed for each escalating dosing period. The actual doses to be administered may be adjusted based on safety, tolerability, and pharmacokinetic data at previous dose levels; these dose adjustments may involve either an increase or a decrease in the planned dose for both Cohorts 1 and 2
  Interventions: Drug: GSK3179106; Drug: Placebo
- Cohort 2 (Experimental): Cohort 2 will proceed after completion of the treatment periods in Cohort 1. Subjects assigned to Cohort 2 will participate in up to 4 dosing periods which include up to 2 escalating doses and placebo in Periods 1 and 2, and a pilot food effect in Periods 3 and 4. A review of safety and tolerability will occur prior to administration of the next dose level and the same procedure will be followed for each escalating dosing period. The actual doses to be administered may be adjusted based on safety, tolerability, and pharmacokinetic data at previous dose levels; these dose adjustments may involve either an increase or a decrease in the planned dose for both Cohorts 1 and 2
  Interventions: Drug: GSK3179106; Drug: Placebo

INTERVENTIONS:
Drug: GSK3179106 — GSK3179106 will be provided as white to slightly colored round or oblong tablet for oral administration with unit dose strength of 5 mg, 25 mg and 100 mg
Drug: Placebo — Placebo will be provided as white to slightly colored round or oblong tablet for oral administration with unit dose strength to match actives across all strengths

SUMMARY:
GSK3179106 is a potent and relatively selective inhibitor of RET kinase which has been designed to be a safe and effective therapy for irritable bowel syndrome (IBS) patients .

This is a randomized, double-blind (sponsor unblind), placebo-controlled, dose escalating, four period, single-dose crossover, first time in human study to assess the safety, tolerability and pharmacokinetics of GSK3179106 in normal healthy subjects.

The study will be composed of 2 cohorts, each having screening (21 days prior to first dose of study drug), Treatment, and follow-up periods (7-10 days after their last dose [Day 1 of dosing period 4]). The Treatment period will include 4 dosing periods. Subjects will participate in either Cohort 1 or Cohort 2. The total duration of the study for each subject will be approximately 10 weeks. A sufficient number of healthy subjects will be screened to enrol 16 subjects who complete the planned study procedures. Each dosing period will be staggered so that only 2 of the 8 subjects will be administered study drug initially. Once 24 hours (h) have elapsed, and provided there are no safety concerns, the remainder of subjects scheduled for that dosing period may be dosed. A review of safety and tolerability will occur prior to administration of the next dose level. This same procedure will be followed for each escalating dosing period. Subjects assigned to Cohort 1 will participate in 1 placebo and 3 dose escalating periods. Subjects assigned to Cohort 2 will participate in up to 4 dosing periods which include up to 2 escalating doses and placebo in Periods 1 and 2, and a pilot food effect in Periods 3 and 4. Within each cohort, subjects will return for their next scheduled dosing period approximately 14 days after administration of the study drug during the prior dosing period. Cohort 2 will proceed after completion of the treatment periods in Cohort 1. Each subject will be enrolled in only one cohort. The planned dose range is 10 milligram (mg) to 200 mg in Cohort 1. The actual doses to be administered may be adjusted based on safety, tolerability, and pharmacokinetic data at previous dose levels; these dose adjustments may involve either an increase or a decrease in the planned dose for both Cohorts 1 and 2. There are no formal hypotheses being tested in this study.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 55 years of age inclusive, at the time of signing the informed consent.
* Healthy as determined by the investigator based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameter(s) which is/are not specifically listed in the inclusion or exclusion criteria, outside the reference range for the population being studied may be included only if the investigator, in consultation with the medical monitor, agree and document that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* History of regular bowel habits.
* Male or Female Males: Male subjects with female partners of child bearing potential must comply with the following contraception requirements from the time of first dose of study medication until at least five half-lives of study medication after the last dose of study medication.

  1. Vasectomy with documentation of azoospermia.
  2. Male condom plus partner use of one of the contraceptive options below:

Contraceptive subdermal implant, Intrauterine device or intrauterine system, Oral Contraceptive, either combined or progestogen alone Injectable progestogen, Contraceptive vaginal ring.

This is an all-inclusive list of those methods that meet the following GlaxoSmithKline (GSK) definition of highly effective: having a failure rate of less than 1 percentage (%) per year when used consistently and correctly and, when applicable, in accordance with the product label. For non-product methods (e.g., male sterility), the investigator determines what is consistent and correct use.

The investigator is responsible for ensuring that subjects understand how to properly use these methods of contraception.

Females: A female subject is eligible to participate if she is of non-reproductive potential defined as: Pre-menopausal females with one of the following:

Documented tubal ligation Documented hysteroscopic tubal occlusion procedure with follow-up confirmation of bilateral tubal occlusion Hysterectomy Documented Bilateral Oophorectomy Postmenopausal defined as 12 months of spontaneous amenorrhea in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) and estradiol levels consistent with menopause (refer to laboratory reference ranges for confirmatory levels). Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the highly effective contraception methods if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrolment.

* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the consent form and in this protocol.

Exclusion Criteria:

* Alanine Transferase (ALT) and bilirubin >1.5x upper limit of normal (ULN) (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Previous diagnosis of IBS.
* Estimated Glomerular Filtration Rate <60 milliliters per minute 1.73 square meter (mL/min/1.73m^2).
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* History of gastroesophageal reflux disease (GERD), dyspepsia, gastrointestinal (GI) bleeding, GI surgery that could affect motility
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
* A positive pre-study drug/alcohol screen.
* A positive test for human immunodeficiency virus (HIV) antibody.
* History of regular alcohol consumption within 6 months of the study defined as: an average weekly intake of >14 standard drinks. One standard drink is equivalent to 10 grams (g) of alcohol: 285 ml of beer, 100 ml of wine or 30 ml of 40% alcohol by volume distilled spirits.
* Current smoker or use of nicotine containing products within the past 3 months or unable to abstain from smoking tobacco or the use of nicotine-containing products while on study.
* Unable to refrain from consumption of red wine, seville oranges, grapefruit or grapefruit juice and/or pummelos, exotic citrus fruits, grapefruit hybrids or fruit juices from 1 day prior to the first dose of study drug on Day 1 of each dosing period, until completion of the last PK blood sample time point for that dose period.
* Corrected QT interval to Fridericia's formula (QTcF) >450 milliseconds (msec)
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Unable to refrain from the use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication for each dosing period until Day 4 of each dosing period, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety. Paracetamol (<=2 grams per day) is acceptable.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than 4 investigational medicinal products within 12 months prior to the first dosing day
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2015-11-26 (Actual); Primary Completion 2016-03-18 (Actual); Study Completion 2016-03-18 (Actual)

PRIMARY OUTCOMES:
Number of subjects with adverse events (AE) and clinical observations as a measure of safety | Up to 10 weeks in each cohort
  An AE is any untoward medical occurrence in a subject or clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Assessment of physical examination findings as a measure of safety | Screening, Day-1 and at follow-up (up to 10 weeks) in each cohort
  Physical examination will include the assessment of the cardiovascular, respiratory, gastrointestinal and neurological systems. A brief physical examination will be conducted at follow-up visit which include, at a minimum assessments of the lungs, cardiovascular system, and abdomen (liver and spleen). Height and weight will also be measured and recorded (height will only be recorded at screening assessment).
Safety as assessed by 12-lead electrocardiogram (ECG) | Up to 10 weeks in each cohort
  Triplicate 12-lead ECGs will be obtained at each time point during the study using an ECG machine that automatically calculates the heart rate and measures PR, QRS, QT, and corrected QT interval (QTc).
Safety as assessed by systolic and diastolic blood pressure measurements | Up to 10 weeks in each cohort
  Three readings of systolic and diastolic pressure will be taken at each time point and the average will be calculated electronically
Safety as assessed by temperature measurements | Up to 10 weeks in each cohort
  Temperature measurements will be taken at Screening, Day-1 and pre-dose in each treatment period. For all other vital sign time points if clinically indicated
Safety as assessed by pulse rate measurements | Up to 10 weeks in each cohort
  Three readings of systolic and diastolic pressure will be taken at each time point and the average will be calculated electronically
Composite of clinical laboratory assessments as a measure of safety includes hematology, clinical chemistry and urinalysis | Up to 10 weeks in each cohort
  Clinical safety laboratory assessments include hematology, clinical chemistry, urinalysis and additional parameters
Bristol Stool Form Scale | Up to Day 4 in each cohort
  The Bristol Stool Form Scale describes 7 types of stool and will be used by the subject to monitor the changes in defecation pattern during the study

SECONDARY OUTCOMES:
Area under the plasma concentration-time curve (AUC) from zero to time t (AUC [0-t]) of GSK3179106 administered under fasting condition | Day 1 Pre-dose and 0.5 h, 1 h, 1.5 h, 2 h, 2.5 h, 3 h, 4 h, 5 h, 6 h, 8 h, 12 h, 18 h, 24 h, 36 h, 48 h, 60 h and 72 h postdose in each treatment period of cohort 1
  PK parameters under fasting conditions
AUC from zero to infinity (AUC [0-infinity]) of GSK3179106 administered under fasting condition | Day 1 Pre-dose and 0.5 h, 1 h, 1.5 h, 2 h, 2.5 h, 3 h, 4 h, 5 h, 6 h, 8 h, 12 h, 18 h, 24 h, 36 h, 48 h, 60 h and 72 h post-dose in each treatment period of cohort 1
  PK parameters under fasting conditions
AUC from zero to 24 h (AUC [0-24 h]) of GSK3179106 administered under fasting condition | Day 1 Pre-dose and 0.5 h, 1 h, 1.5 h, 2 h, 2.5 h, 3 h, 4 h, 5 h, 6 h, 8 h, 12 h, 18 h, 24 h, 36 h, 48 h, 60 h and 72 h post-dose in each treatment period of cohort 1
  PK parameters under fasting conditions
Maximum observed plasma concentration (Cmax) of escalating single oral doses of GSK3179106 administered under fasting conditions | Day 1 Pre-dose and 0.5 h, 1 h, 1.5 h, 2 h, 2.5 h, 3 h, 4 h, 5 h, 6 h, 8 h, 12 h, 18 h, 24 h, 36 h, 48 h, 60 h and 72 h post-dose in each treatment period of cohort 1
  PK parameters under fasting conditions
Time to maximum observed plasma concentration (tmax) of GSK3179106 administered under fasting condition | Day 1 Pre-dose and 0.5 h, 1 h, 1.5 h, 2 h, 2.5 h, 3 h, 4 h, 5 h, 6 h, 8 h, 12 h, 18 h, 24 h, 36 h, 48 h, 60 h and 72 h post-dose in each treatment period of cohort 1
  PK parameters under fasting conditions
Apparent terminal phase half-life (t1/2) of GSK3179106 administered under fasting condition | Day 1 Pre-dose and 0.5 h, 1 h, 1.5 h, 2 h, 2.5 h, 3 h, 4 h, 5 h, 6 h, 8 h, 12 h, 18 h, 24 h, 36 h, 48 h, 60 h and 72 h post-dose in each treatment period of cohort 1
  PK parameters under fasting conditions
Clearance (CL/F) of GSK3179106 administered under fasting condition | Day 1 Pre-dose and 0.5 h, 1 h, 1.5 h, 2 h, 2.5 h, 3 h, 4 h, 5 h, 6 h, 8 h, 12 h, 18 h, 24 h, 36 h, 48 h, 60 h and 72 h post-dose in each treatment period of cohort 1
  PK parameters under fasting conditions
Volume of distribution (V/F) of GSK3179106 administered under fasting condition | Day 1 Pre-dose and 0.5 h, 1 h, 1.5 h, 2 h, 2.5 h, 3 h, 4 h, 5 h, 6 h, 8 h, 12 h, 18 h, 24 h, 36 h, 48 h, 60 h and 72 h post-dose in each treatment period of cohort 1
  PK parameters under fasting conditions
Absorption rate constant (Ka) of GSK3179106 administered under fasting condition | Day 1 Pre-dose and 0.5 h, 1 h, 1.5 h, 2 h, 2.5 h, 3 h, 4 h, 5 h, 6 h, 8 h, 12 h, 18 h, 24 h, 36 h, 48 h, 60 h and 72 h post-dose in each treatment period of cohort 1
  PK parameters under fasting conditions
Area under the plasma concentration-time curve (AUC) from zero to time t (AUC [0-t]) of GSK3179106 administered under fasting and fed condition | Day 1 Pre-dose and 0.5 h, 1 h, 1.5 h, 2 h, 2.5 h, 3 h, 4 h, 5 h, 6 h, 8 h, 12 h, 18 h, 24 h, 36 h, 48 h, 60 h and 72 h post-dose in each treatment period of cohort 2
  PK parameters under fasting and fed conditions
AUC from zero to infinity (AUC [0-infinity]) of GSK3179106 administered under fasting condition fasting and fed condition | Day 1 Pre-dose and 0.5 h, 1 h, 1.5 h, 2 h, 2.5 h, 3 h, 4 h, 5 h, 6 h, 8 h, 12 h, 18 h, 24 h, 36 h, 48 h, 60 h and 72 h post-dose in each treatment period of cohort 2
  PK parameters under fasting and fed conditions
AUC from zero to 24 h (AUC [0-24 h]) of GSK3179106 administered under fasting condition fasting and fed condition | Day 1 Pre-dose and 0.5 h, 1 h, 1.5 h, 2 h, 2.5 h, 3 h, 4 h, 5 h, 6 h, 8 h, 12 h, 18 h, 24 h, 36 h, 48 h, 60 h and 72 h post-dose in each treatment period of cohort 2
  PK parameters under fasting and fed conditions
Maximum observed plasma concentration (Cmax) of escalating single oral doses of GSK3179106 administered under fasting and fed condition | Day 1 Pre-dose and 0.5 h, 1 h, 1.5 h, 2 h, 2.5 h, 3 h, 4 h, 5 h, 6 h, 8 h, 12 h, 18 h, 24 h, 36 h, 48 h, 60 h and 72 h post-dose in each treatment period of cohort 2
  PK parameters under fasting and fed conditions
Time to maximum observed plasma concentration (tmax) of GSK3179106 administered under fasting and fed condition | Day 1 Pre-dose and 0.5 h, 1 h, 1.5 h, 2 h, 2.5 h, 3 h, 4 h, 5 h, 6 h, 8 h, 12 h, 18 h, 24 h, 36 h, 48 h, 60 h and 72 h post-dose in each treatment period of cohort 2
  PK parameters under fasting and fed conditions
Apparent terminal phase half-life (t1/2) of GSK3179106 administered under fasting and fed condition | Day 1 Pre-dose and 0.5 h, 1 h, 1.5 h, 2 h, 2.5 h, 3 h, 4 h, 5 h, 6 h, 8 h, 12 h, 18 h, 24 h, 36 h, 48 h, 60 h and 72 h post-dose in each treatment period of cohort 2
  PK parameters under fasting and fed conditions
Clearance (CL/F) of GSK3179106 administered under fasting and fed condition | Day 1 Pre-dose and 0.5 h, 1 h, 1.5 h, 2 h, 2.5 h, 3 h, 4 h, 5 h, 6 h, 8 h, 12 h, 18 h, 24 h, 36 h, 48 h, 60 h and 72 h post-dose in each treatment period of cohort 2
  PK parameters under fasting and fed conditions
Volume of distribution (V/F) of GSK3179106 administered under fasting and fed condition | Day 1 Pre-dose and 0.5 h, 1 h, 1.5 h, 2 h, 2.5 h, 3 h, 4 h, 5 h, 6 h, 8 h, 12 h, 18 h, 24 h, 36 h, 48 h, 60 h and 72 h post-dose in each treatment period of cohort 2
  PK parameters under fasting and fed conditions
Absorption rate constant (Ka) of GSK3179106 administered under fasting and fed condition | Day 1 Pre-dose and 0.5 h, 1 h, 1.5 h, 2 h, 2.5 h, 3 h, 4 h, 5 h, 6 h, 8 h, 12 h, 18 h, 24 h, 36 h, 48 h, 60 h and 72 h post-dose in each treatment period of cohort 2
  PK parameters under fasting and fed conditions

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Adelaide, South Australia, Australia

REFERENCES:
- [Derived] Cooper M, O'Connor-Semmes R, Reedy BA, Hacquoil K, Gorycki P, Pannullo K, Verticelli A, Shakib S. First-in-Human Studies for a Selective RET Tyrosine Kinase Inhibitor, GSK3179106, to Investigate the Safety, Tolerability, and Pharmacokinetics in Healthy Volunteers. Clin Pharmacol Drug Dev. 2019 Feb;8(2):234-245. doi: 10.1002/cpdd.600. Epub 2018 Sep 13. PMID 30277655
- See also: Results for study 204729 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/204729?search=study&b'search_terms=204729'#rs